CLINICAL TRIAL: NCT07393659
Title: A Phase 3b, Open-label, Multicenter, Continued Access Study for Participants Transitioning From ViiV Healthcare Sponsored or ViiV Healthcare Collaborative Parent Studies for HIV Treatment
Brief Title: A Continued Access Study for Participants Transitioning From ViiV Healthcare-sponsored or ViiV Healthcare-collaborative Parent Studies for HIV Treatment
Acronym: PATH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300269
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus (HIV); Open label; Continued access
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continued Access Group (Experimental): Participants with HIV-1 who received the study intervention and completed the protocol-defined treatment period in ViiV Healthcare-sponsored or ViiV Healthcare-collaborative parent studies (2020-001029-30, 2020-001426-57), and who continue to receive the study intervention from their respective parent study.
  Interventions: Drug: Fostemsavir; Drug: Dolutegravir (DTG)/ Lamivudine (3TC)

INTERVENTIONS:
Drug: Fostemsavir — Participants receive oral tablets with the dosages depending on the weight of the participants.
Drug: Dolutegravir (DTG)/ Lamivudine (3TC) — Participants receive oral tablets with the dosages depending on the weight of the participants.

SUMMARY:
The purpose of this study is to provide continued access to the study treatment for participants from previous ViiV Healthcare studies who are still benefiting from it and do not have local access after completing the parent study. This continued access will also allow further collection of safety data. Eligible participants are those who completed a ViiV Healthcare-sponsored or collaborative parent study and are currently experiencing clinical benefit. The Sponsor will periodically review the study to consider other treatment access options.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in this study only if all the following criteria apply:

* Investigator confirmation of the participant's continued clinical benefit from the parent study intervention and the participant's completion of the protocol-defined treatment period in the parent study. The Investigator should ensure that the participant is still eligible for the parent study (i.e., have not met parent study discontinuation/ withdrawal criteria).
* Participants or legally authorized representative (LAR) who are willing and able to comply with all scheduled visits, treatment plan, and other study procedures as outlined in the applicable appendix and determined by the Investigator.
* Participant or LAR is able and willing to provide signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and this protocol. Where applicable, participants must provide written assent.

Exclusion Criteria:

Participants are excluded from participating in this study if the following criterion applies:

• Any reason that, in the opinion of the Investigator or Sponsor, precludes the participant's inclusion in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2026-05-08 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who discontinue the study intervention and the reason for discontinuation | Throughout the study period (from rollover visit at Day 1 until the end of study/withdrawal visit)
Number of participants with serious adverse events (SAE) | Throughout the study period (from rollover visit at Day 1 until the end of study /withdrawal visit)
  A SAE is defined as any untoward medical occurrence that, at any dose, results in results in death, is life- threatening, requires inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, abnormal pregnancy outcomes or a suspected transmission of any infectious agent via an authorized medicinal product.
Number of participants with adverse events of special interest (AESI) | Throughout the study period (from rollover visit at Day 1 until the end of study /withdrawal visit)
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AESI is defined as an AE of a scientific and medical concern specific to the study intervention, which may require further investigation in order to characterize and understand it.

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf